CLINICAL TRIAL: NCT00287599
Title: Rapid Identification of Key Pathogens in Wound Infection by Molecular Means
Status: Completed | Type: Observational
Sponsor: Brentwood Biomedical Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: W81XWHO510134
Record Dates: First submitted 2006-02-03; First posted 2006-02-07 (Estimated); Last update posted 2012-02-08 (Estimated); Status verified 2012-02

CONDITIONS: Postoperative Wound Infection; Traumatic Wound Infection; Closed Soft Tissue Abscess
Keywords: Surgical wound infections; Real-time PCR; Rapid identification of bacteria; Cloning; 16S rRNA sequencing
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Pus and tissue specimens
Oversight: Data Monitoring Committee: No

SUMMARY:
The military is subject to traumatic wounds of various types and severity. Such wounds are predisposed to infection because they 1) tend to be extensive and deep, 2) may affect areas of normal carriage of potentially pathogenic bacteria in the gastrointestinal tract, upper respiratory tract, and the female genital tract, 3) typically produce tissue damage, 4) may introduce foreign bodies, 5) may interfere with local blood supply, 6) tend to produce ischemia, edema and hemorrhage, 7) may be complicated by fractures or burns and 8) may lead to shock and overwhelming of the body's systemic defenses. It will not always be possible in the military setting to cleanse and debride the wound promptly and effectively or to promptly provide surgery in the event of damage to vital structures. In the active military setting, the probability of wound infection following trauma is relatively high. In the absence of rapid identification of infecting flora and provision of information on antimicrobial susceptibility, clinicians must resort to empiric therapy rather than a tailored therapy. There is a tendency to use one of the top available agents that would likely be active against the vast majority of bacteria. This leads to increases in antimicrobial resistance, an important problem.

The investigators hypothesize that the use of molecular biology techniques will provide identification of the microorganisms responsible for wound infection more rapidly and accurately. The investigators will evaluate real-time PCR (polymerase chain reaction) technique under this proposal. This procedure can be applied directly to material from the wound without need for first growing the organisms. It can be used to define the total flora of the wound within five hours. The investigators will first develop primers and probes that will detect the various bacteria anticipated in a given wound in a certain location. These primers and probes will be used in real-time PCR for rapid and accurate identification of the wound flora. The information obtained with real-time PCR is quantitative so that one may judge the relative importance of different isolates. The investigators will also use another molecular approach, 16S rRNA gene cloning, and conventional cultures; these will provide further information about the flora of various wounds. Definitive identification of anaerobes can be provided quickly and that, along with information on usual antimicrobial susceptibility patterns, can be life-saving or shorten the course of the infection considerably.

DETAILED DESCRIPTION:
Background: Wound infections are typically mixed, with both anaerobic and non-anaerobic bacteria present and there are usually more anaerobes than aerobes (for example, in perforated or gangrenous appendicitis, we have found an average of 9 anaerobes and 3 aerobes). Many clinical laboratories do limited anaerobic bacteriology, using commercial kits based on inadequate phenotypic characteristics and inaccurate taxonomy. As a result, physicians and surgeons must treat wound infections empirically and tend to use drugs active against the most resistant anaerobes which leads to increased resistance to antimicrobials. Molecular techniques now available permit accurate and rapid characterization of microorganisms, both aerobic and anaerobic.

Objective/Hypothesis: The use of molecular biology techniques will provide identification of the microorganisms responsible for wound infection both more rapidly and more accurately. The current conventional method of culture and identification by phenotypic testing is slow and inaccurate.

Specific Aims: 1) Develop a rapid identification method, to include quantitation, for important wound pathogens, 2) Analyze bacterial flora of wound infection by molecular means and by conventional culturing; both tissue biopsies and pus will be studied by both methodologies, 3) Determine the incidence and significance of the so-called "uncultivable" flora.

Study Design: We will study 50 postoperative and traumatic wound infections and 50 closed soft tissue abscesses in intravenous drug abusers annually, from a general surgical service at Olive View County Hospital, affiliated with UCLA and the VA Medical Center West Los Angeles, in collaboration with Dr. Robert Bennion. Whenever possible, we will obtain tissue biopsies from the active edge of the wound for processing, along with pus from the wound.

We will develop species-specific primers/probes for organisms that are encountered in different types of wound infections based on information about the flora of wound infection obtained from previous studies by our group and others and supplemented with primers/probes made from cultural isolates not previously encountered. The primers and probes will be used in a high-throughput procedure (real-time PCR) that permits rapid identification and quantitation of organisms. The entire procedure, including both DNA extraction and real-time PCR, can be completed within 5 hours for one sample. Multiple samples can be done concurrently. While it may be necessary to start therapy empirically, it will be possible to change to more appropriate antimicrobial agents when the bacteriologic data becomes available in 5 hours. Concurrently, we will utilize another molecular approach, 16S rRNA gene cloning, to analyze the total flora of the sample. We will first amplify 16S rRNA genes using universal (all bacteria) primers by PCR of DNA extracted from the sample. Then, a clone library will be constructed in E. coli and all clones will be studied by 16S rDNA sequencing of ~1500 base pairs. This permits detection of organisms called "uncultivable", as well as organisms that can be cultured successfully. Any "uncultivable" organisms that are encountered frequently may be important; therefore, we will develop primers and probes for their rapid identification and we will use a variety of techniques to attempt to cultivate these (we have done this successfully in a few cases already). At the same time as the molecular approaches are being done, we will use conventional cultural processing. The cultural approach will provide organisms for additional study (especially for antimicrobial susceptibility testing) and will serve as the current standard for comparison with the newer molecular approaches. Culture will be done semiquantitatively and identification will be done by 16S rDNA sequencing supplemented by phenotypic testing as indicated. The cultural approach typically takes several days to isolate the organisms in pure culture.

The two molecular approaches will be compared with the conventional cultural approach in terms of organisms detected; each specimen will be studied by all techniques, for comparative purposes.

Relevance: The speed of the various identification schemes indicated above shows clearly that we would be able to provide accurate, quantitative identification (more accurate than by the conventional cultural approach) a great deal sooner than has been possible in the past. This should lead to much earlier application of the most appropriate therapy and minimize empiric use of our most powerful agents. This is likely to result in improved clinical outcome, less chance for antimicrobial resistance, and cost savings as well. It will provide us with a much more accurate picture of the infecting flora of various surgical wounds and the antimicrobial susceptibility pattern of these organisms. We will learn whether, as in burn wound infections, quantitative study of tissue biopsies will provide a better picture of the true infecting flora than conventional wound cultures. We will learn whether "uncultivable" bacteria (which actually make up the greatest percentage of the indigenous flora of the bowel and the upper respiratory tract) are important clinically or not. Finally, we will develop a more complete set of primers/probes to improve the molecular approach.

ELIGIBILITY:
Inclusion Criteria:

* active postoperative or traumatic wound infection
* soft tissue abscess

Exclusion Criteria:

* no active infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2006-10; Primary Completion 2009-09 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sydney M Finegold, MD, Principal Investigator — VA Medical Center-West Los Angeles
Locations (2):
- United States (2):
  - Sydney Finegold, Los Angeles, California
  - Robert S Bennion MD, Sylmar, California